CLINICAL TRIAL: NCT03317977
Title: Translating an Efficacious Illness Management Intervention for Youth With Poorly Controlled Asthma to Real World Settings
Brief Title: Translating an Efficacious Illness Management Intervention for Youth With Asthma
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Wayne State University (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Principal Investigator, Deborah Ellis, Ph.D., Professor of Family Medicine and Public Health Sciences, Wayne State University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 071217MP4E; R01HL138633-01A1 (NIH)
Record Dates: First submitted 2017-10-18; First posted 2017-10-23 (Actual); Results first posted 2024-04-04 (Actual); Last update posted 2024-04-04 (Actual); Status verified 2024-04

CONDITIONS: Asthma in Children
Keywords: Asthma management, adolescents

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Reach for Control (Experimental): Reach For Control is a multi-component, home-based family therapy that targets the multiple causes of poor adolescent asthma management across individual, family and community systems.
  Interventions: Behavioral: Reach for Control
- Michigan MATCH (Active Comparator): Program endorsed by the State of Michigan for treatment of poorly controlled asthma.
  Interventions: Behavioral: MATCH

INTERVENTIONS:
Behavioral: Reach for Control — In Phase 1 (weeks 1-4), the CHW conducts an initial intake and then completes a comprehensive functional analysis (FA) of behavior to determine the causes of poor asthma management for each youth regarding asthma management. In Phase 2 (weeks 5-20) is a treatment phase and consists of a combination of mandatory cognitive-behavioral skills training (CBST) modules (received by all families) and flexible CBST modules chosen and individualized based on the results of the Phase 1 FA. This includes but not limited to In-vivo Asthma Skills Training, Improving Family Communication and Behavioral Contracting. Phase 3 (weeks 21-24) involves termination planning and relapse prevention
  Other Names: RFC
  Arms: Reach for Control
Behavioral: MATCH — Managing Asthma Through Case Management in Home (MATCH) is the current intervention provided by WCHAP to youth with poorly controlled asthma and their families.
  Arms: Michigan MATCH

SUMMARY:
The propose of the study is to test the effectiveness of Reach for Control (RFC) as compared to Michigan MATCH to improve asthma symptoms, asthma management and lung functioning and to decrease ED visits and admissions for youth with poorly controlled asthma when integrated into hospital emergency departments and delivered by community health workers. The study is a hybrid implementation-effectiveness design and will test RFC for use in real world, public healthcare settings.

DETAILED DESCRIPTION:
The study was conducted in the emergency department at Children's Hospital of Michigan; CHM). 170 adolescents with poorly controlled asthma and their primary caregivers will be enrolled. Prior to the COVID-19 pandemic, families were randomly assigned to six months of home-based family treatment consisting of either RFC or Michigan MATCH , a model program endorsed by the State of Michigan for treatment of poorly controlled asthma. Subsequently, all intervention content in both arms was delivered by telehealth. Treatment content of RFC consists of weekly sessions focusing on asthma education, asthma management skills, improving home-school community for asthma, access to care and case management. MATCH includes asthma education but is less intensive and does not focus on family management skills. Treatment was provided by community health workers (CHWs) employed by a community agency providing MATCH as their standard of care. Consent and data collection was completed at baseline with additional data collection visits at 6, 12 and 18 months after baseline. Data collection was completed by project research assistants and consists of questionnaires and interviews with the adolescent and parent to assess asthma management, asthma symptoms and hospital utilization. The data analyses were intent-to-treat, meaning that all randomized participants are included regardless of the intervention dose received. Trial data were analyzed using linear mixed effect models.

ELIGIBILITY:
Inclusion Criteria:

Adolescent/Parent:

1. Child aged 12 years, 0 months to 16 years, 11 months
2. Moderate to severe persistent asthma
3. Child seen in the CHM emergency department for treatment of asthma exacerbation
4. Child has experienced 2 or more ED visits and/ or inpatient admissions in prior 12 months (i.e. poorly controlled asthma)
5. Parent/ legal guardian willing to participate in home-based family treatment
6. Child and family resides within 20 miles of CHM (allows for home-based data collection and intervention)

Exclusion Criteria:

Adolescent/Parent:

1. Child is currently in an out-of-home placement
2. Schizophrenia or other psychosis on the part of the youth or parent
3. Current suicidality or homicidality on the part of the youth or parent
4. Cognitive impairment or learning disability that prevents comprehension of research measures on the part of parent or youth

Ages: 12 Years to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 75 (Actual)
Dates: Start 2018-02-01 (Actual); Primary Completion 2023-08-08 (Actual); Study Completion 2023-08-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Deborah A Ellis, Ph.D, Principal Investigator — Wayne State University
Locations (1):
- Children's Hospital of Michigan, Detroit, Michigan, United States

IPD SHARING:
Plan to Share IPD: Yes
Data will be made available at the end of the study through presentations at scientific conferences and publications in peer-reviewed scientific journals. All final peer-reviewed manuscripts that result from the study will be submitted to PubMed Central. In addition, final dataset from the trial will be shared. Identifiers will be removed from the data prior to any release of the dataset.
Time Frame: Indefinitely
Access Criteria: In light of the sensitive nature of the treatment data contained in the data set, as well as the participation of children, data and associated documentation will be made available to users only under a specific data-sharing agreement that provides for: (1) a commitment to using the data only for research purposes and not to identify any individual participant; (2) a commitment to securing the data using appropriate computer technology; and (3) a commitment to destroying the data after analyses are completed. Furthermore, audiotaped session recordings will not be shared, as these include voice identifiers and it is not possible to de-identify the recordings; costs of transcription of sessions given their length and number are beyond the scope of the study.

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited from the emergency department of a large urban tertiary care pediatric hospital
Groups:
- Michigan MATCH: Managing Asthma Through Case Management in Home (MATCH) is the current intervention provided by WCHAP to youth with poorly controlled asthma and their families.The program has been endorsed by the State of Michigan as a model program for poorly controlled asthma.
Period: Overall Study
Arm/Group | Reach for Control | Michigan MATCH
Started | 36 | 39
Completed | 31 | 35
Not Completed | 5 | 4

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Reach for Control | Michigan MATCH | Total
Number analyzed (Participants) | 36 | 38 | 74
Age, Continuous [Mean (Standard Deviation); unit: years] | 14.5 (1.3) | 14.4 (1.4) | 14.4 (1.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 19 | 20 | 39
  Male | 17 | 18 | 35
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Black | 35 | 35 | 70
  White | 1 | 3 | 4
Region of Enrollment [Number; unit: participants]
  United States | 36 | 38 | 74
Asthma Control Test [Mean (Standard Deviation); unit: units on a scale] — The measure is a self-report questionnaire that consists of five items: activity limitation, shortness of breath, night-time awakenings due to asthma symptoms, use of quick- relief medication and a global rating of asthma control. Items are rated on a 1-5 scale over the past four weeks, with higher scores indicating better control over asthma symptoms. The total score ranges from 5 to 25 with higher scores indicating better control over asthma symptoms.
  units on a scale | 18.9 (3.8) | 18.5 (4.4) | 18.7 (4.1)

OUTCOME MEASURES:

1. Primary Outcome: Number of Emergency Department Visits
Description: Emergency department visits will be obtained from electronic medical records
Time Frame: Change from Baseline at 6 months, 12 months, and 18 months
Population: All randomized participants were analyzed with the exception of study removals
Measure: Mean (Standard Deviation); unit: Count of ED visits in prior six months
Arm/Group | Reach for Control | Michigan MATCH
Number analyzed (Participants) | 36 | 38
Count of ED visits in prior six months
  Baseline | 0.67 (0.79) | 0.68 (0.70)
  6-month change | 0.28 (0.45) | 0.50 (1.18)
  12-month change | 0.14 (0.42) | 0.26 (0.55)
  18-month change | 0.08 (0.28) | 0.03 (0.16)
Statistical Analysis 1: Comparison: Michigan MATCH; Test type: Superiority; p = 0.43, Mixed Models Analysis

2. Secondary Outcome: Family Asthma Management System Scale
Description: Identifies family strengths and weaknesses in the management of pediatric asthma across a variety of domains. This is a semi-structured interview that is rated on seven to nine 9-point subscales with higher scores indicating better management. The rating manual provides elaboration and brief examples at key anchor points for each rating scale. A FAMSS summary score is computed for each family by taking a mean across all subscales.
Time Frame: Change from Baseline at 6 months, change from Baseline at 12 months and change from Baseline at 18 months
Reporting Status: Not Posted

3. Secondary Outcome: Asthma Symptom Frequency
Description: Self report assessing wheezing, nighttime symptoms, speech limitations and activity limitations.
Time Frame: Change from Baseline at 6 months, change from Baseline at 12 months and change from Baseline at 18 months
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: 1 year
Arm/Group | Reach for Control | Michigan MATCH
All-Cause Mortality (participants affected / at risk) | 0/36 | 0/38
Serious Adverse Events (participants affected / at risk) | 4/36 | 7/38
Other Adverse Events (participants affected / at risk) | 18/36 | 20/38
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Reach for Control (N=36) | Michigan MATCH (N=38)
Hospitalization (Respiratory, thoracic and mediastinal disorders) | 4 (6) | 5 (8) — Hospitalization for an asthma related event.
New Family Problem (Social circumstances) | 0 (0) | 1 (1)
New Health Problem (General disorders) | 0 (0) | 1 (1) — New health problem not related to asthma.
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Reach for Control (N=36) | Michigan MATCH (N=38)
New Family Problem (Social circumstances) | 5 (5) | 6 (8)
New Health Problem (General disorders) | 9 (13) | 5 (6)
New Problem with Parent-Child Relations (Social circumstances) | 2 (2) | 5 (5)
New Psychiatric Problem (Psychiatric disorders) | 3 (3) | 2 (2)
New School-Related Problem (Social circumstances) | 3 (3) | 2 (2)
Worsening Family Problem (Social circumstances) | 2 (2) | 1 (1)
Worsening Health Problem (General disorders) | 11 (15) | 14 (37)
Worsening Psychiatric Problem (Psychiatric disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2024-02-12): https://cdn.clinicaltrials.gov/large-docs/77/NCT03317977/Prot_SAP_000.pdf
  • Informed Consent Form (2023-03-28): https://cdn.clinicaltrials.gov/large-docs/77/NCT03317977/ICF_001.pdf